CLINICAL TRIAL: NCT04172363
Title: Clinical Relevance of the Antimicrobial Resistance Testing in the Treatment of Chronic Wounds With Antiseptics
Acronym: AntiSeptic
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left site
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-169
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Decubiti; Chronic Wounds; Acute Wounds
MeSH Terms: conditions — Pressure Ulcer | interventions — octenidine and phenoxyethanol drug combination

STUDY DESIGN:
Intervention Model Description: This is monocentric, prospective, controlled, open, randomized, 2-armed interventional pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Octenisept will be used as standard care antiseptic for dressing change
- Resistance testing (Experimental): Patients will be first tested on resistance to Octenisept and Serasept and will receive the appropriate antiseptic after reviewing the results
  Interventions: Drug: Octenisept and Serasept

INTERVENTIONS:
Drug: Octenisept and Serasept — Swab probes of wounds will be taken upon study inclusion and analysed for resistance on Octenisept and Serasept. If the patient indicates resistance on one of the antiseptics, he/she will receive the other antiseptic for wound dressings
  Arms: Resistance testing

SUMMARY:
The study objective is to improve the current and local standard antiseptic treatment by adjusting the antiseptic agent to the antimicrobial resistance testing result, accordingly. Currently, resistance testing will only be performed for the treatment with antibiotics.

DETAILED DESCRIPTION:
Complications like bacterial wound colonization and infections in wound treatment are still a serious problem. Several therapy approaches are available to treat these complications, e.g. surgical wound debridement, antimicrobial therapy that can be divided into a local and a systemic antisepsis.

The local antisepsis (the local utilization of antiseptics directly to the wound) is in many ways advantageous to the systemic antisepsis (orally or intravenously administered antibiotics): e. g. the direct contact of the antiseptic to the bacteria at the site of infection whereas antibiotics may not sufficiently reach the wound due to limited blood perfusion of wounds; growing utilization of systemic antisepsis also leads to an increasing number of resistant bacteria worldwide. To the concerns of many specialists, the first pan-resistant bacterial strain which is resistant to all available antibiotics including colistin was recently published.

In future, the role of local antisepsis therefore becomes more important in the antimicrobial treatment. Luckily, resistances of local antiseptics occur slowly due to the chemical and structural characteristics of antiseptics but even resistances of bacteria to antiseptics were reported. Unlike the antimicrobial resistance testing for antibiotics that is done in the clinical routine, such testing is not a standard procedure for antiseptics for no obvious reason. The utilization of antiseptics is determined by the availability of products provided within the institution and preferences of the clinician. Thus, it is unknown whether the chosen antiseptic has any bactericidal effect on the confirmed bacteria.

University Hospital RWTH Aachen Wound Care only uses polyhexanide and octenisept. Iodine-containing preparations are explicitly not desired.Improvement (bacteria reduction, acceleration of wound healing) of the local antiseptic therapy by adapting the antiseptic to the results of antimicrobial resistance testing. Antimicrobial resistance testing has so far only been used to adapt systemic antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Decubitus OR secondary healing acute and chronic wounds
3. Positively tested wound swab for bacteria (incl. multi-resistant bacteria)
4. Patient is capable of understanding the nature, significance and consequence of the clinical trial
5. Given written consent
6. Women of child bearing potential (WOCBP) who apply appropriate methods of contraception throughout the duration of the study

Exclusion Criteria:

1. Occlusive dressing (e.g. VAC) or Negative Pressure Wound Therapy (NPWT)
2. Pregnant or lactating women
3. Known allergies against investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-22 (Estimated); Primary Completion 2021-05-22 (Estimated); Study Completion 2021-05-22 (Estimated)

PRIMARY OUTCOMES:
Change in bacteria rate | up to 12 months
  determination of the relative proportion of isolates to the total flora in the wound

SECONDARY OUTCOMES:
Incidence of wound related adverse events | up to 12 months
  review of medical charts
Change in Pressure Ulcers: Scale for Healing (PUSH) score | up to 12 months
  score 0-17; 17=big and severe wound
Change in Bates-Jensen Score | up to 12 months
  Score 13-65; 13-20=minimal severity class; 41-65 extreme severity class
Laboratory Parameters - Change in C-reactive protein (CRP) | up to 12 months
  mg/L
Laboratory Parameters - Change in Leukocytes | up to 12 months
  10⁹/L or /nL
Laboratory Parameters - Change in hemoglobin | up to 12 months
  g/dl
Laboratory Parameters - Change in hematokrit | up to 12 months
Laboratory Parameters - Change in creatinine | up to 12 months
  µmol/L or mg/dl
Laboratory Parameters - Change in glomerular filtration rate (GFR) | up to 12 months
  ml/min/1,73m^2
Laboratory Parameters - Change in Uric acid | up to 12 months
  mg/dl
Laboratory Parameters - Change in glutamic-pyruvic transaminase (GPT) | up to 12 months
  IU/L
Laboratory Parameters - Change in Glutamat-Oxalacetat- Transaminase (GOT) | up to 12 months
  IU/L
Laboratory Parameters - Change in Glucose | up to 12 months
  mmil/L or mg/dl
Hospital length of stay | up to 12 months
  from study inclusion until hospital discharge
Rate of antibiotics used | up to 12 months
  chart review
Length of bed confinement | up to 12 months
  chart review

CONTACTS AND LOCATIONS:
Overall Officials: Christian Stoppe, Prof., Principal Investigator — Aachen University Hospital
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No